CLINICAL TRIAL: NCT03807193
Title: Self-selected or Predetermined Internet-based Cognitive Behavior Therapy for Generalized Anxiety Disorder With Weekly Support or Support on Demand: A Factorial Treatment Study
Brief Title: Self-selected or Predetermined Internet-based Treatment for Generalized Anxiety Disorder With Different Types of Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: worry factorial
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: Worry
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: A factorial design with four cells:
  Cell one: Predetermined treatment program with weekly support Cell two: Predetermined treatment program with support on demand Cell three: Self-selected treatment program with weekly support Cell four: Self-selected treatment program with support on demand
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fixed treatment, weekly support (Experimental): Receives a predetermined treatment program and have weekly support.
  Interventions: Behavioral: Predetermined treatment; Behavioral: Weekly support
- Fixed treatment, support on demand (Experimental): Receives a predetermined treatment program and have access to support on demand.
  Interventions: Behavioral: Predetermined treatment; Behavioral: Support on demand
- Selected treatment, weekly support (Experimental): Select their own treatment material and have weekly support.
  Interventions: Behavioral: Self-selected treatment; Behavioral: Weekly support
- Selected treatment, support on demand (Experimental): Select their own treatment material and have access to support on demand.
  Interventions: Behavioral: Self-selected treatment; Behavioral: Support on demand

INTERVENTIONS:
Behavioral: Self-selected treatment — The participants will select their own treatment material with the help of a written manual. The interventions possible to choose are all interventions used in standard cognitive behavior therapy for anxiety and depression.
  Arms: Selected treatment, support on demand; Selected treatment, weekly support
Behavioral: Predetermined treatment — The participants will be given a treatment program designed to address worry and generalized anxiety disorder. The program are based on newer forms of cognitive behavior therapy and include mindfulness and acceptance.
  Arms: Fixed treatment, support on demand; Fixed treatment, weekly support
Behavioral: Weekly support — The participants will have scheduled weekly support, once a week, during the treatment. The support till be delivered by students in clinical psychology.
  Arms: Fixed treatment, weekly support; Selected treatment, weekly support
Behavioral: Support on demand — The participants will have support if and when they ask for it by themselves. If asked for the support will be delivered by students in clinical psychology.
  Arms: Fixed treatment, support on demand; Selected treatment, support on demand

SUMMARY:
This study evaluates two types of internet-based treatments for generalized anxiety disorder and two types of support. The treatments are a predetermined program for generalized anxiety disorder and a self-selected treatment. The different types of support are either a weekly contact trough a secure message system or support on demand.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is characterize by and excessive and uncontrollable worry that is present more days than not. The disorder is best described as a chronic condition with periods with more or less symptoms. The disorder is highly disabling with low quality of life for the individual and is associated with and high costs for society. Previous studies on internet-based cognitive behavior therapy for GAD has shown positive effects but there are still room for improvement.

The aim of this study is to evaluate two different internet-based treatments as well as two types of support through the use of a factorial design. The participants will be recruited trough advertising. After registration on the study's website the potential participants will be asked to answer screening questionnaires and demographic data for an initial screening. Those meeting inclusion criteria will be contacted for a diagnostic interview based Mini-International Neuropsychiatric Interview (M.I.N.I.). If meeting the study's inclusion criteria and not the exclusion criteria the participant will be included in the study and randomized to one of the four arms. The four arms are: Predetermined treatment program with weekly support, Predetermined treatment program with support on demand, Self-selected treatment with weekly support, Self-selected treatment with support on demand.

The predetermined treatment program is designed for treatment of worry and generalized anxiety disorder. It is based on newer forms of cognitive behavior therapy and includes mindfulness and acceptance. In the self-selected treatment the participants will select treatment interventions with the help of a manual and encouraged to choose interventions that they feel address their specific problems. The interventions that will be available are all based on standard cognitive behavior therapy techniques. The weekly support will be scheduled and delivered by clinical psychology students under supervision. This contact will be based on reports from the participants on the weeks work with the program and exercises. The support on demand will be also be delivered by clinical psychology students under supervision. This support takes place if and when the participant ask for support. Treatment will be 8 weeks long and both treatments will be delivered through the same platform. Contact with the participants will be trough written messages on a secure platform.

After the eight weeks of treatment the participants will be asked to answer the same measures as before the treatment as well as questions regarding how they experience the treatment. Follow up data will be collected at later points.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* fulfilling criteria for generalized anxiety syndrome
* 45 points or more on PSWQ
* Able to read and write in Swedish
* Have daily access to a computer and internet

Exclusion Criteria:

* Alcohol or substance abuse
* Acute suicidal
* Ongoing psychological treatment
* Ongoing medication for anxiety or depression that is planned to be adjusted during the time of the treatment given in the study
* Complex psychiatric illness that highly disabling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Penn State Worry Questionnaire (PSWQ) | Baseline, 8 weeks, 24 months and 36 months after treatment
  Measures symptoms severity of worry. 16 items, with score range 16-80. Higher score indicates worse symptoms

SECONDARY OUTCOMES:
Change from baseline in Generalized Anxiety Disorder Questionnaire IV (GAD-Q-IV) | Baseline, 8 weeks, 24 months and 36 months after treatment
  Designed to capture the criteria for generalized anxiety disorder according to diagnostic and statistical manual of mental disorders (DSM), 9 items with score range 0-12. Higher scores indicate greater symptom severity
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | baseline and weekly during 8 weeks treatment. 24 months and 36 months after treatment
  Screening measure for worry and anxiety symptoms. 7 items, score range 0-21. Higher scores indicate greater symptom severity
Change from baseline in Beck Anxiety Inventory (BAI) | Baseline, 8 weeks, 24 months and 36 months after treatment
  Measure of anxiety symptoms. 21 items with score range 0-63. Higher scores indicate greater symptom severity
Change from baseline in Patient Health Questionnaire (PHQ-9) | baseline and weekly during 8 weeks treatment. 24 months and 36 months after treatment
  Screening measure for depressive symptoms. 9 items with score range 0-27. Higher scores indicate greater symptom severity
Beck Depression II Inventory (BDI-II) | Baseline, 8 weeks, 24 months and 36 months after treatment
  Measure of severity of depressive symptoms. 21 items with score range 0-63. Higher scores indicate greater symptom severity
Acceptance and Action Questionnaire II (AAQ-II) | Baseline, 8 weeks, 24 months and 36 months after treatment
  Measure of psychological flexibility. 7 items with score range 7-49 with higher scores indicate lower psychological flexibility
Brunnsviken Brief Quality of life scale (BBQ) | Baseline, 8 weeks, 24 months and 36 months after treatment
  12 items, measures the quality of life. 12 items with score 0-96. Higher score indicate higher quality of life
General self-efficacy scale | Baseline, 8 weeks, 24 months and 36 months after treatment
  Measure of percieved self-efficay. 10 items rated on a four-point Likert scale. Score range 10-40 with a higher score indicating a higher percieved self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linköpings universitet, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided